CLINICAL TRIAL: NCT02778308
Title: Randomized Controlled Trial Comparing Adjuvant Chemotherapy Vs. no Chemotherapy for Patients With Carcinoma of Gallbladder Undergoing Curative Resection.
Brief Title: Adjuvant Chemotherapy vs no Chemotherapy for Patients With GallBllader Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Institute of Postgraduate Medical Education and Research (Other Government)
Responsible Party: Principal Investigator, Sundeep Singh Saluja, Associate Professor, Govind Ballabh Pant Institute of Postgraduate Medical Education and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FI/IEC/MAMC(32)/4/2012/239
Record Dates: First submitted 2016-03-06; First posted 2016-05-19 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Gallbladder Cancer
Keywords: Gallbladder cancer, adjuvant chemotherapy, gemcitabine
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy group (Active Comparator): 6 cycles of Gemcitabine + Cisplatin as per the following schedule Injection Gemcitabine 1 gm/kgm2 intravenous over 30 min Day1 and Day8 Injection Cisplatin 70 mg/m2 intravenous on Day1
  Interventions: Drug: Gemcitabine + Cisplatin
- control group (No Intervention): follow up

INTERVENTIONS:
Drug: Gemcitabine + Cisplatin — Day 1 and day 8 Gemcitabine Day 1 cisplatin
  Other Names: GemCis
  Arms: chemotherapy group

SUMMARY:
Carcinoma of the gallbladder is the commonest malignancy of the biliary tract. Higher incidence has been noted in Chile, Mexico and Southwest American Indians.[1] It is the third most common malignancy in India.[2] The disease may mimic benign disease in presentation.Up to 1/3rd of patients may present with jaundice but of these only 7% will be resectable.[4] With aggressive surgical resection, actuarial 5 year survival of 83% for stage II disease and 63% for stage III have been reported.[5] Treatment of choice is complete surgical resection.

The role of chemotherapy and radiotherapy is not very well documented in treatment of gallbladder cancer. Because of the propensity of gallbladder carcinoma to spread to regional lymph nodes at an early stage and the high rate of loco regional recurrence, adjuvant chemotherapy or chemo-radiotherapy seems a rational therapeutic option. Gemcitabine with or without Cisplatin has been increasingly used. In a recent paper Gemcitabine with Cisplatin was found to be more effective than gemcitabine alone and provides definite survival advantage and progression free survival.[6] An earlier randomized trial done to assess the efficacy of the adjuvant chemotherapy for the pancreato-biliary cancer reported improvement in disease free and overall 5 year survival.[7] But this study has included patients with suboptimal resection and all pancreato-biliary malignancy.

In view of these observations this study is being designed to assess the efficacy of the chemotherapy in the adjuvant setting in gallbladder cancer patients who have undergone curative resections.

DETAILED DESCRIPTION:
Carcinoma of the gallbladder is the commonest malignancy of the biliary tract. United states has an incidence of 1/100000.Higher incidence has been noted in Chile, Mexico and Southwest American Indians. It is the third most common malignancy in India. The disease may mimic benign disease in presentation. Now 78-85% of the cases may be detected preoperatively with radiological imaging. 1-3% of the carcinoma of the gall bladder may be detected incidentally. Up to 1/3rd of patients may present with jaundice but of these only 7% will be resectable. With aggressive surgical resection, actuarial 5 year survival of 83% for stage II disease and 63% for stage III have been reported. Treatment of choice is complete surgical resection.

The role of chemotherapy and radiotherapy is not very well documented in treatment of gallbladder cancer. Because of the propensity of gallbladder carcinoma to spread to regional lymph nodes at an early stage and the high rate of loco regional recurrence, adjuvant chemotherapy or chemo-radiotherapy seems a rational therapeutic option. The chemotherapies are based on 5 Fluorouracil with or without radiotherapy. Gemcitabine with or without Cisplatin has been increasingly used. In a recent paper Gemcitabine with Cisplatin was found to be more effective than gemcitabine alone and provides definite survival advantage and progression free survival. An earlier randomized trial done to assess the efficacy of the adjuvant chemotherapy for the pancreato-biliary cancer reported improvement in disease free and overall 5 year survival. But this study has included patients with suboptimal resection and all pancreato-biliary malignancy.

In view of these observations this study is being designed to assess the efficacy of the chemotherapy in the adjuvant setting in gallbladder cancer patients who have undergone curative resections.

ELIGIBILITY:
Inclusion Criteria:

1. T1b and above adenocarcinoma of gall bladder
2. Patients undergoing curative resection
3. Incidentally diagnosed carcinoma who have undergone curative completion radical cholecystectomy

Exclusion Criteria:

1. T1a tumors
2. Patients with metastatic disease
3. Patients unfit to undergo chemotherapy
4. Patients unwilling to undergo the trial
5. Patients with double cancers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival | From date of randomization until the date of first documented recurrence, assessed up to 100 months.
  Defined as the time interval between the date of randomization and the date of disease recurrence.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  Defined as the time interval between the date of randomization and death from disease or unrelated cause
Blood and lymphatic system Adverse events | till 6 weeks after last cycle
  As per CTCAE version 5 criteria
Gastrointestinal system Adverse events | Till 6 weeks after last cycle
  As per CTCAE version 5 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pramod K Mishra, Phd, Study Chair — GIPMER; Kishore Singh, MD, Study Director — Lok Nayak Hospital
Locations (1):
- GIPMER, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Perkin DM, Whelan SL, Ferlay J, Raymond L, Young J. Cancer incidence in five continents. Vol VII, Lyon, France: International Agency for Research on Cancer Scientific Publication No. 143, 1997.
- [Background] Shukla VK, Khandelwal C, Roy SK, Vaidya MP. Primary carcinoma of the gall bladder: a review of a 16-year period at the University Hospital. J Surg Oncol. 1985 Jan;28(1):32-5. doi: 10.1002/jso.2930280109. PMID 3968886
- [Background] Hamrick RE Jr, Liner FJ, Hastings PR, Cohn I Jr. Primary carcinoma of the gallbladder. Ann Surg. 1982 Mar;195(3):270-3. doi: 10.1097/00000658-198203000-00005. PMID 7059239
- [Background] Hawkins WG, DeMatteo RP, Jarnagin WR, Ben-Porat L, Blumgart LH, Fong Y. Jaundice predicts advanced disease and early mortality in patients with gallbladder cancer. Ann Surg Oncol. 2004 Mar;11(3):310-5. doi: 10.1245/aso.2004.03.011. PMID 14993027
- [Background] Bartlett DL, Fong Y, Fortner JG, Brennan MF, Blumgart LH. Long-term results after resection for gallbladder cancer. Implications for staging and management. Ann Surg. 1996 Nov;224(5):639-46. doi: 10.1097/00000658-199611000-00008. PMID 8916879
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Takada T, Amano H, Yasuda H, Nimura Y, Matsushiro T, Kato H, Nagakawa T, Nakayama T; Study Group of Surgical Adjuvant Therapy for Carcinomas of the Pancreas and Biliary Tract. Is postoperative adjuvant chemotherapy useful for gallbladder carcinoma? A phase III multicenter prospective randomized controlled trial in patients with resected pancreaticobiliary carcinoma. Cancer. 2002 Oct 15;95(8):1685-95. doi: 10.1002/cncr.10831. PMID 12365016
- [Derived] Saluja SS, Nekarakanti PK, Mishra PK, Srivastava A, Singh K. Prospective Randomized Controlled Trial Comparing Adjuvant Chemotherapy vs. No Chemotherapy for Patients with Carcinoma of Gallbladder Undergoing Curative Resection. J Gastrointest Surg. 2022 Feb;26(2):398-407. doi: 10.1007/s11605-021-05143-6. Epub 2021 Sep 20. PMID 34545545